CLINICAL TRIAL: NCT05028959
Title: Menstrual Cycle, Amenorrhea and Contraception in Elite Female Athletes: Impact on Performance, Health and the Athlete's Biological Passport
Brief Title: Hormonal Status, Performance and Health in Elite Female Athlete
Acronym: FEMMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Paris-Saclay-Assistance publique des hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Emmanuelle Duron, Head of Geriatry, Principal investigator, Université Paris-Saclay-Assistance publique des hôpitaux de Paris
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FEM-2020
Record Dates: First submitted 2021-06-21; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: female elite athlete; menstrual phase; amenorrhea; hormonal contraception; performance; health; Athlete Biological Passport
MeSH Terms: conditions — Amenorrhea

STUDY DESIGN:
Intervention Model Description: 2 groups : female athletes and leisure sports women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Female athletes (Experimental): highly trained subjects
  Interventions: Other: Multidisciplinary monitoring of healthy women
- Leisure sport women (Experimental): recreational sportswomen practicing regular physical activity
  Interventions: Other: Multidisciplinary monitoring of healthy women

INTERVENTIONS:
Other: Multidisciplinary monitoring of healthy women — Multidisciplinary monitoring

SUMMARY:
The repercussions of the hormonal status of high-level sportswomen on their performance and health as well as on the Athlete's Biological Passport (ABP) have been little studied and remain poorly known. The investigators therefore propose to contribute to the improvement of current knowledge by determining, thanks to the implementation of a multidisciplinary monitoring, with the use of various tests and matrices, in female elite athletes and recreational athletes (control group):

* 1) the impact of cycle phase, absence of cycle or contraceptive use on physical and psychological performance, health as well as on ABP;
* 2) the potential confounding effects of the athlete's environment
* 3) correlations between the different matrices analyzed

DETAILED DESCRIPTION:
Volunteers to be studied: 80 healthy female subjects (16 to 30 years old), divided into 2 groups:

Group 1: 60 athletes, from different sports disciplines, in amenorrhea, with menstrual cycle or taking contraceptives

Group 2: 20 leisure sports subjects with menstrual cycle or taking contraceptives

Following the oral and written information of the project, the subjects have a minimum of 15 days of reflection before signing the written consent form. They will have the possibility, at any time, to voluntarily interrupt the study without having to justify themselves.

Investigations to be performed:

1. Annual complete clinical examination :
2. "Out-of-competition" follow-up, time frame 6 months

   * medical, nutritional and respiratory monitoring
   * biological monitoring
   * psychological monitoring
   * performance monitoring
3. Non-invasive "in-competition" monitoring, only for Group 1, once in a year on the day before/after a major competition:

   * biological monitoring
   * psychological monitoring
   * performance monitoring (interview)

ELIGIBILITY:
Inclusion Criteria:

* Group 1: high-level athletes (qualified for national/international championships and/or training at least 15 hours/week)
* Group 2: recreational athletes who practice a regular physical activity

Exclusion Criteria:

* Participation in another trial
* History of cardiac pathology
* High blood pressure
* History of ulcers and other gastrointestinal disorders
* Myasthenia
* Renal insufficiency
* Person not affiliated or not benefiting from a social security system

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline weight | 6 months
  in kg, by impedancemeter
Change from baseline fat and lean mass | 6 months
  in kg, by impedancemeter
Change from baseline height | 6 months
  in cm, by height gauge
Change from baseline sex and stress hormones | 6 months
  concentration of oestradiol, progesterone, testosterone, DHEA, cortisol, LH and FSH in mol/L
Change from baseline food intake | 6 months
  food intake questionnaire to complete over 3 days, expressed in kcal/day
Change from baseline metabolic parameters | 6 months
  concentration of blood glucose, blood lactate, lipid profile, insulin, GH, IGF1, T3, IgA, PRL and leptin in mol/L
Change from baseline respiratory parameters | 6 months
  measure of FEV1 (forced expiratory volume in 1 second), expressed in % of vital capacity
Change from baseline inflammatory parameters | 6 months
  concentration of cytokines (TNF-alpha, IL-6) in mol/L
Change from baseline executive function | 6 months
  assessed by instability via static and dynamic postures (eyes open/closed) on platform
Change from baseline visual-spatial processing | 6 months
  3 D mental rotation test, assessed by scores: range from 0 - 24, with 24 representing a perfect total score
Change from baseline attention and working memory | 6 months
  Stroop Color Word Task, assessed by scores : range of interference from -15 - +15, with higher scores representing decreased selective attention
Change from baseline performance monitoring | 6 months
  field performance test, performance expressed in time
Change from baseline Athlete Biological Passport (Group 2) | 6 months
  assessed by analysis of the standardized parameters of the Athlete Biological Passport (WADA)
Change from baseline affects (Group 2) | 6 months
  Positive Affect and Negative Affect Schedule (PANAS), assessed by scores. Positive Affect Score: range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: range from 10 - 50, with lower scores representing lower levels of negative affect.
Change from baseline anxiety (Group 2) | 6 months
  Spielberger State-Trait Anxiety Inventory, assessed by scores: range from 20 - 80, with higher scores representing higher anxiety
Change from baseline Athlete Biological Passport (Group 1) | 8 months
  assessed by analysis of the standardized parameters of the Athlete Biological Passport (WADA)
Change from baseline affects (Group 1) | 8 months
  Positive Affect and Negative Affect Schedule (PANAS), assessed by scores. Positive Affect Score: range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: range from 10 - 50, with lower scores representing lower levels of negative affect.
Change from baseline anxiety (Group 1) | 8 months
  Spielberger State-Trait Anxiety Inventory, assessed by scores: range from 20 - 80, with higher scores representing higher anxiety
Interview (Group 1) | 8 months
  Self-confrontation interview for questioning the action

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackerman KE, Singhal V, Baskaran C, Slattery M, Campoverde Reyes KJ, Toth A, Eddy KT, Bouxsein ML, Lee H, Klibanski A, Misra M. Oestrogen replacement improves bone mineral density in oligo-amenorrhoeic athletes: a randomised clinical trial. Br J Sports Med. 2019 Feb;53(4):229-236. doi: 10.1136/bjsports-2018-099723. Epub 2018 Oct 9. PMID 30301734
- [Background] Crewther BT, Cook CJ. The salivary testosterone response to a chance-determined contest is associated with face-gazing behaviours in athletic women. Horm Behav. 2018 Jul;103:107-110. doi: 10.1016/j.yhbeh.2018.06.011. Epub 2018 Jul 2. PMID 29953884
- [Background] Casey E, Reese M, Okafor E, Chun D, Gagnon C, Nigl F, Dhaher YY. Influence of Menstrual Cycle and Oral Contraceptive Phase on Spinal Excitability. PM R. 2016 Sep;8(9):860-8. doi: 10.1016/j.pmrj.2016.01.013. Epub 2016 Feb 10. PMID 26872589
- [Background] Cornelli U, Belcaro G, Cesarone MR, Finco A. Analysis of oxidative stress during the menstrual cycle. Reprod Biol Endocrinol. 2013 Aug 2;11:74. doi: 10.1186/1477-7827-11-74. PMID 23915183
- [Background] Eklund E, Berglund B, Labrie F, Carlstrom K, Ekstrom L, Hirschberg AL. Serum androgen profile and physical performance in women Olympic athletes. Br J Sports Med. 2017 Sep;51(17):1301-1308. doi: 10.1136/bjsports-2017-097582. Epub 2017 Jun 23. PMID 28646101
- [Background] Emami F, Kordi Yoosefinejad A, Motealleh A. Comparison of static and dynamic balance during early follicular and ovulation phases in healthy women, using simple, clinical tests: a cross sectional study. Gynecol Endocrinol. 2019 Mar;35(3):257-260. doi: 10.1080/09513590.2018.1519788. Epub 2018 Oct 23. PMID 30350735
- [Background] Hausmann M, Slabbekoorn D, Van Goozen SH, Cohen-Kettenis PT, Gunturkun O. Sex hormones affect spatial abilities during the menstrual cycle. Behav Neurosci. 2000 Dec;114(6):1245-50. doi: 10.1037//0735-7044.114.6.1245. PMID 11142657
- [Background] Julian R, Hecksteden A, Fullagar HH, Meyer T. The effects of menstrual cycle phase on physical performance in female soccer players. PLoS One. 2017 Mar 13;12(3):e0173951. doi: 10.1371/journal.pone.0173951. eCollection 2017. PMID 28288203
- [Background] Kishali NF, Imamoglu O, Katkat D, Atan T, Akyol P. Effects of menstrual cycle on sports performance. Int J Neurosci. 2006 Dec;116(12):1549-63. doi: 10.1080/00207450600675217. PMID 17145688
- [Background] Kluft C, Leuven JA, Helmerhorst FM, Krans HM. Pro-inflammatory effects of oestrogens during use of oral contraceptives and hormone replacement treatment. Vascul Pharmacol. 2002 Aug;39(3):149-54. doi: 10.1016/s1537-1891(02)00304-x. PMID 12616983
- [Background] Langdeau JB, Day A, Turcotte H, Boulet LP. Gender differences in the prevalence of airway hyperresponsiveness and asthma in athletes. Respir Med. 2009 Mar;103(3):401-6. doi: 10.1016/j.rmed.2008.09.023. Epub 2008 Nov 21. PMID 19027280
- [Background] Lebrun CM, Petit MA, McKenzie DC, Taunton JE, Prior JC. Decreased maximal aerobic capacity with use of a triphasic oral contraceptive in highly active women: a randomised controlled trial. Br J Sports Med. 2003 Aug;37(4):315-20. doi: 10.1136/bjsm.37.4.315. PMID 12893716
- [Background] Nose-Ogura S, Yoshino O, Dohi M, Kigawa M, Harada M, Hiraike O, Onda T, Osuga Y, Fujii T, Saito S. Risk factors of stress fractures due to the female athlete triad: Differences in teens and twenties. Scand J Med Sci Sports. 2019 Oct;29(10):1501-1510. doi: 10.1111/sms.13464. Epub 2019 Jun 9. PMID 31100189
- [Background] Otaka M, Chen SM, Zhu Y, Tsai YS, Tseng CY, Fogt DL, Lim BH, Huang CY, Kuo CH. Does ovulation affect performance in tennis players? BMJ Open Sport Exerc Med. 2018 Jan 27;4(1):e000305. doi: 10.1136/bmjsem-2017-000305. eCollection 2018. PMID 29464104
- [Background] Schaumberg MA, Jenkins DG, Janse DE Jonge XA, Emmerton LM, Skinner TL. Oral Contraceptive Use Dampens Physiological Adaptations to Sprint Interval Training. Med Sci Sports Exerc. 2017 Apr;49(4):717-727. doi: 10.1249/MSS.0000000000001171. PMID 27898641